CLINICAL TRIAL: NCT01388712
Title: The Assessment of Lactobacillus Reuteri Efficacy, Provided With Forlax, as Treatment of Incurable Constipation in Children 3-7 Years. Double Blind, Placebo-controlled, Randomized and Multicenter Trial
Brief Title: Lactobacillus Reuteri in Children With Constipation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Memorial Health Institute, Poland (Other)
Responsible Party: Principal Investigator, JAROSLAW KIERKUS, Ph.D., Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CZDGA23.01.2011
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Functional Constipation
Keywords: Probiotics; constipation; children
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Probiotics (Active Comparator): Lactobacillus reuteri DSM 17938
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — Patients, who met inclusion criteria, will receive following medicaments during 8 weeks: Lactobacillus reuteri DSM 17938 in form of chewing (one tablets containing 10^8CFU).
  Arms: Probiotics
Dietary Supplement: Placebo — Patients, who met inclusion criteria, will receive an identical to probiotic looking and tasting placebo.
  Arms: Placebo

SUMMARY:
The most common cause of children chronic constipation is functional disorders. Functional constipation is diagnosed after excluding organic causes of constipation (anatomical, neurological, endocrinological) and identification of two symptoms defined by the Rome III criteria. There could be low number of bowel movements (below three times a week), defecation pain, fecal incontinence (once a week), stool consistency or occurrence of large diameter stools. The treatment is change of diet, defecation training and application of laxatives.

The probiotics are defined as living microorganisms, which provided in a proper doses should result in beneficial effect on a host health. The assessment of its characteristic is related to strain of bacteria affiliation.

Taking into the consideration that patients with constipation may experience microflora intestine disorders, using the probiotics can have the positive impact on process of treating this disease. The additional reason for using the probiotics during the constipation treatment is an influence of probiotics on movement of the alimentary canal.

In spite of proved effectiveness of some probiotics' strains further research are required, because clinical significance is ambiguous and the effect is confirmed among patients with short medical history. That's way the further analysis of probiotic Lactobacillus reuteri DSM 17938, which was successful treatment method of chronic constipation amongst children (infants) should be performed.

The primary aim of the study is the assessment of Lactobacillus reuteri DSM 17938 efficacy, provided with macrogol (Forlax), as treatment of constipation in 3-7 years old children. The baseline of estimation is the frequency comparison of bowel movement in children belonging into two groups: Lactobacillus reuteri treatment and placebo.

The secondary aim of the study is the assessment of frequency the additional symptoms connected with defecation disorders: such as: number of pain episodes during defecation, the intensity of pain, number of hard stools, number of fecal incontinence per week, number of macrogol (Forlax) pockets used.

The investigators believe that constipation treatment (laxatives- macrogol) with Lactobacillus reuteri has better efficacy that the same treatment without Lactobacillus reuteri in 3-7 years old children with medical history of chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-7 years old
* Occurrence less than three bowel movement per week
* Medical history from at least two months]
* Ineffective laxative treatment at least two months
* The parents approval for child participation in the study and for the treatment

Exclusion Criteria:

* Well-known, organic cause of constipation (i.e. hypothyroidism, Hirschprung disease, cystis fibrosis)
* Anatomic defects of the alimentary canal
* The surgery of the alimentary canal in the past
* Treatment of antibiotics/probiotics during last two weeks before start of the study

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-04 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Number of bowel movement per week, without fecal incontinence | 12 weeks

SECONDARY OUTCOMES:
The number of bowel movements per week | 12 weeks
  Other secondary items are: the number of pain episodes during defecation per week, the number of hard stools, the number of fecal incontinence per week, the number of patients who have to change amount of drug or use of enema.
The number of pain episodes during defecation per week, | 12 weeks
The number of hard stools | 12 weeks
The number of fecal incontinence per week | 12 weeks
The number of patients who have to change amount of drug | 12 weeks
The number of patients who have to change use of enema. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Kierkus, Ph.D., Study Chair — Children's Memorial Health Institute, Poland; Agnieszka Wegner, M.D., Principal Investigator — Children's Memorial Health Institute, Poland
Locations (1):
- ChildrensMHIPoland, Warsaw, Poland